CLINICAL TRIAL: NCT06905340
Title: Nociception Level Index-Guided Intraoperative Opioids in Patients With a Combination of General and Regional Anesthesia
Brief Title: Guiding Opioid Administration by Nociception Level Index (NOL) in Patients With Regional Anesthesia
Acronym: NORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TEMP522873-BO-ff
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Nociceptive Pain; Pain, Postoperative; Analgesia, Postoperative; Anesthesia Recovery Period; Opioid Use
Keywords: General anesthesia; Regional anesthesia; Analgesia Monitoring; Opioids
MeSH Terms: conditions — Nociceptive Pain; Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blinded to the three primary endpoints (postoperative pain level in the PACU, postoperative opioid consumption in the PACU, and postoperative opioid consumption in the first 24 hours after the operation). Patients are blinded to group allocation. Postoperative outcome parameters are assessed by members of the study team. These outcome assessors are blinded to the group assignment.
  During the operation, the attending anesthesiologists cannot be blinded to group allocation because the study involves intervention during the intraoperative treatment. As such, the study is only single-blinded regarding the intraoperative secondary endpoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NOL (Nociception Level Index) (Experimental): Opioid administration (sufentanil) guided by the Nociception Level Index (NOL) derived from photoplethysmography, galvanic skin conductance, and the measurement of skin temperature performed by the device PMD-200 Nociception Monitor from the manufacturer Medasense Biometrics Ltd, Ramat Yishai, Israel. Included in the monitoring system is software that continuously calculates the NOL from normalized heart rate variability, pulse plethysmographic amplitude, skin conductance, and skin temperature derived from a finger sensor. The numerical index ranges from 0 (low sympathetic tone) to 100 (high sympathetic tone). A NOL score between 10 and 25 has been proposed as the target range based on which to guide opioid analgesics dosage. 5 µg sufentanil will be administered if the NOL score exceeds 25 for more than 60 seconds. The sufentanil boluses may be repeated to keep NOL between 10-25 accordingly.
  Interventions: Procedure: NOL (Nociception Level Index)
- Control (Active Comparator): Opioid administration (sufentanil) based on standard clinical practice where attending anesthesiologists are advised to administer 5 µg sufentanil if signs of inadequate anesthesia are present. Given adequate hypnosis (BIS 40-60), these signs include hypertension (MAP>120% of baseline or >100mmHg), tachycardia (HR>120% of baseline or >90/min), somatic arousal (coughing, chewing, grimacing) and somatic response (purposeful movement). The patient-specific baseline is defined as the average of three consecutive post-induction, pre-surgery MAP and HF values. The time elapsed between 5µg doses of sufentanil is up to the anesthesiologist's discretion.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Procedure: NOL (Nociception Level Index) — Elective surgery in patients having trauma and orthopedic surgery with a combination of general and regional anesthesia. Opioid titration is guided by NOL during general anesthesia in the experimental arm.
  Arms: NOL (Nociception Level Index)
Other: Control (Standard treatment) — Opioid administration (sufentanil) guided according to standard clinical practice of the attending anesthesiologist
  Arms: Control

SUMMARY:
General anesthesia consists of a combination of hypnotic drugs to achieve unconsciousness and opioid analgesics to ensure antinociception. An alternative approach to the intraoperative administration of high-potency opioids to achieve antinociception during surgery is combining general anesthesia with regional anesthesia. Modern general anesthesia aims to avoid an overdose of opioid analgesics and reduce side effects of opioid administration. Quality and safety of general anesthesia are of major clinical importance and can be improved by adjusting the opioid analgesics to the optimal individual dose needed.

In current clinical practice, opioid dosage is usually determined by clinical judgment. However, different monitoring devices estimating the effect of nociception during unconsciousness have become commercially available. One of the most recent commercially available nociception indices is the Nociception Level Index (NOL). Until today, there is conflicting evidence on whether guiding sufentanil administration by NOL monitoring, which is the intended use of the nociception index, affects postoperative pain level in the postanesthesia care unit (PACU), the amount of postoperatively administered opioids, and the quality of postoperative recovery in patients with a combination of general and regional anesthesia. This study aims to investigate the clinical performance of intraoperative NOL monitoring and determine whether guiding sufentanil administration by NOL monitoring - compared to routine care - reduces either postoperative pain level in the PACU, postoperative opioid consumption in the PACU or postoperative opioid consumption in the first 24 hours after the operation in patients having trauma and orthopedic surgery with combined general and regional anesthesia.

DETAILED DESCRIPTION:
Modern general anesthesia aims to treat nociception induced by surgical stimulation while avoiding an overdose of opioid analgesics and reducing side effects of opioid administration.

Underdosing of opioids during surgery can lead to nociception with increased sympathetic tone, elevated levels of stress hormones, unintended patient movement as well as increased postoperative pain. On the other hand, overdosing of opioids can lead to negative side effects such as nausea and vomiting, arterial hypotension, immunosuppression, prolonged recovery times, postoperative delirium and an increase in postoperative pain by opioid-induced hyperalgesia. Anesthesiologists therefore aim to strike the balance between an effective and long-lasting perioperative anesthesia/analgesia, and keeping the intra- and postoperative opioid dosage as high as needed, but as low as possible to reduce adverse effects. An alternative approach to the intraoperative administration of high-potency opioids for achieving antinociception during surgery is combining general anesthesia with regional anesthesia. By combining the two, the anesthesiologists aim to reduce intraoperative and postoperative opioid administration without compromising reflex control of the autonomous nervous system, immobility of the surgical site without patients' defensive movements, a pain-free awakening after surgery and a pain-free postoperative recovery.

Critically, the quality of regional anesthesia cannot be assessed during general anesthesia by the anesthesiologist, and patients cannot express their pain themselves. Therefore, anesthesiologists tend to administer a certain calculated opioid dose during the operation. Whether this calculated opioid administration is essential for a sufficient anesthesia or is an unnecessary overdose cannot be assessed by the anesthesiologist. To this day, there has been no measurement tool that could estimate the effectiveness of regional anesthesia and the absence of nociception during general anesthesia combined with regional anesthesia.

In recent years, different monitoring devices estimating the effect of nociception during unconsciousness have become commercially available. Such monitoring devices should help physicians to choose the right dose of opioid analgesics during general anesthesia with nociception indices. Among those, the Nociception Level Index (NOL) developed by Medasense Biometrics Ltd, Ramat Yishai, Israel is one of the most promising nociception indices regarding a possible improvement of postoperative patient recovery. This commercially available nociception index has been developed for guiding intraoperative sufentanil administration, has received CE certification for the EU area and an approval by the FDA. The NOL is based on the four physiological parameters heart rate variability, pulse plethysmographic amplitude, skin conductance and skin temperature, which are all measured with a non-invasive finger sensor. A proprietary algorithm generates the NOL from the changes in the four parameters over time using a non-linear random forest regression method through machine learning.

The dimensionless index is presented on a scale from 0 (low sympathetic tone) to 100 (high sympathetic tone) caused by nociception during surgery. According to the manufacturer, a value above 25 indicates a clinically relevant nociceptive response to noxious stimuli while a value below 10 during an operation lasting for more than 2 minutes indicates excessively high analgesia.

Nevertheless, the current literature remains inconclusive about the impact of NOL-guided opioid administration. There is conflicting evidence on the anesthesia-related outcome parameters postoperative pain level, intraoperatively and postoperatively administered amount of opioids, postoperative short-term recovery, and long-term outcome. No study has yet evaluated whether one may estimate the effectiveness of regional anesthesia during general anesthesia by monitoring the intraoperative nociception with the NOL. If the NOL was able to assess nociception, NOL-guided opioid administration could possibly reduce postoperative pain level in the PACU, postoperative opioid consumption in the PACU and postoperative opioid consumption in the first 24 hours after the operation on the ward. Such a reduction of the perioperative opioid dose would constitute a clinically important benefit for patients when considering the previously detailed risks of overdosing opioid analgesics as well as the context of perioperatively developed opioid addiction. Nevertheless, it remains unknown whether guiding sufentanil administration by NOL monitoring affects the administered amount of intraoperative and postoperative opioid consumption, immediate postoperative pain in the PACU and the quality of postoperative recovery, which is the intended use of the nociception index, in patients with a combination of general and regional anesthesia.

This prospective, randomized controlled trial aims to investigate the clinical performance of intraoperative NOL monitoring and determine whether guiding sufentanil administration by NOL monitoring - compared to routine care - reduces either postoperative pain level in the PACU, postoperative opioid consumption in the PACU or postoperative opioid consumption in the first 24 hours after the operation in patients undergoing trauma and orthopedic surgery with a combination of general and regional anesthesia. The hypothesis tested in the present study is that in patients having trauma and orthopedic surgery with a combination of general and regional anesthesia, administration of sufentanil guided by NOL monitoring reduces either postoperative pain level in the PACU, postoperative opioid consumption in the PACU or postoperative opioid consumption in the first 24 hours after the operation compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing elective trauma or orthopedic surgery with a combination of general and regional anesthesia

Exclusion Criteria:

* Preexisting therapy with cardiac glycosides or pacemakers
* Cardiac arrhythmia (atrial fibrillation, atrioventricular block > I°)
* Chronic opioid misuse
* Intraoperative treatment with ketamine, beta-adrenergic agonists, or clonidine
* Serious peripheral or cardiac autonomic neuropathy
* Inability to specify the postoperative pain level
* Postoperative treatment in an ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain level in the PACU | 1 day
  Compares the proportion of postoperative pain level (NRS=0 vs. NRS>0) in the postanesthesia care unit (PACU) between the groups.
Postoperative administration of opioids during the PACU stay | 1 day
  Compares the proportion of postoperative administration of opioids during the PACU stay (none vs. any) between the groups.
Postoperative administration of opioids in the first 24 hours after the operation | 2 days
  Compares the proportion of postoperative administration of opioids in the first 24 hours after the operation (none vs. any) between the groups.

SECONDARY OUTCOMES:
Intraoperative sufentanil consumption | 1 day
  Compares intraoperative sufentanil consumption [μg/kg/min] between the groups.
Intraoperative norepinephrine consumption | 1 day
  Compares intraoperative cumulative dose of norepinephrine consumption [μg/kg/min] between the groups.
Time to extubation | 1 day
  Compares the time from end of narcotics to extubation [min] between the groups.
Postoperative nausea and vomiting (PONV) | 1 day
  Compares the incidence of postoperative nausea and vomiting (PONV) (%) between the groups.
PACU stay | 1 day
  Compares the length of stay in the postanesthesia care unit (PACU) (min) between the groups.
Postoperative pain level 24 hours after the operation | 2 days
  Compares the postoperative pain level at rest 24 hours after the operation (NRS 0-10) between the groups.
Quality-of-Recovery QoR-15 Score | 2 days
  Compares the quality of postoperative recovery measured by the Quality-of-Recovery QoR-15 Score (0-120 points) 24 hours after the operation between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Nitzschke, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg Eppendorf, Hamburg, Germany